CLINICAL TRIAL: NCT07210294
Title: The Effect of Press Needle on Body Acupuncture Points and Auricular Acupuncture Points on Functional Dyspepsia
Brief Title: Press Needle on Body Acupuncture Points and Auricular Acupuncture Points on Functional Dyspepsia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Maria Anastasia Darmawan, MD, Indonesia University
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 25-05-0594
Record Dates: First submitted 2025-09-29; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Functional Dyspepsia
MeSH Terms: interventions — Dosage Forms

STUDY DESIGN:
Intervention Model Description: The intervention group received press needles and medication, while the control group received sham press needles and medication.
Who Masked: Participant, Outcomes Assessor
Masking Description: The participants and the outcome asssesors will be blinded to group allocation
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): The press needle and medication
  Interventions: Device: The press needle and medication
- Control Group (Sham Comparator): The sham press needle and medication
  Interventions: Device: The sham press needle and medication

INTERVENTIONS:
Device: The press needle and medication — Press needles using the needle sizes 0.17mm x 0.9mm on auricular acupuncture points (MA-IC6 (Stomach) bilaterally) and the needle sizes 0.20 mm x 1.5mm on body acupuncture points (ST36 bilaterally). After that, apply an adhesive patches on top of the press needle. The press needle is attached for 14 days (on the 7th day the press needle is replaced).
  Medication using proton pump inhibitor drugs
  Arms: Intervention Group
Device: The sham press needle and medication — Sham press needle uses adhesive patches without needles on auricular acupuncture points (MA-IC6 (Stomach) bilateral) and body acupuncture points (ST36 bilateral). The sham press needle is attached for 14 days (on the 7th day the sham press needle is replaced).
  Medication using proton pump inhibitor drugs
  Arms: Control Group

SUMMARY:
The aim of this study was to prove that press needle (PN) and medication are more effective in reducing symptoms and improving quality of life in people with functional dyspepsia compared to sham press needle (Sham PN) and medication.

The main questions this study aims to answer are:

* Does the press needle and medication group reduce symptoms in people with functional dyspepsia as assessed by the Short Form-Leeds Dyspepsia Questionnaire (SF-LDQ) compared to the sham press-needle and medication group on days 7 and 14, compared to before therapy?
* Does the press-needle and medication group improve quality of life in people with functional dyspepsia as assessed by the Short-Form Nepean Dyspepsia Index (SF-NDI) compared to the sham press-needle and medication group on days 7 and 14, compared to before therapy?

A total of 38 participants were randomly allocated into two groups, either PN or Sham PN needle groups

Participants will:

* Receive PN or Sham PN for 14 days and replaced on day 7.
* Complete the SF-LDQ and SF-NDI questionnaires before therapy, on day 7, and day 14.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-59 years
* Patients with functional dyspepsia
* Esophagogastroduodenoscopy (EGD) results show no significant structural abnormalities or no structural abnormalities.
* Willing to participate in the research until completion and sign a letter of consent for medical action (informed consent).

Exclusion Criteria:

* At the acupuncture point location there is inflammation, malignancy, and scar tissue.
* Deformity of the earlobe.
* History of allergies to stainless steel and plaster.
* Medical emergencies, impaired consciousness, pregnancy, history of diabetes mellitus, and history of keloid formation.
* History of digestive tract cancer, history of hepatobiliary cancer, history of chronic kidney failure stage 4 and 5, history of hyperthyroidism or hypothyroidism.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2026-07-06 (Estimated); Study Completion 2026-07-06 (Estimated)

PRIMARY OUTCOMES:
Short-Form Leeds Dyspepsia Questionnaire (SF-LDQ) | Before therapy, day 7, day 14
  Short-Form Leeds Dyspepsia Questionnaire (SF-LDQ) is a questionnaire consisting of 4 questions A and B. The total score ranges from 0 to 32.
Short-Form Nepean Dyspepsia Index (SF-NDI) | Before therapy, day 7, day 14
  Short-Form Nepean Dyspepsia Index (SF-NDI) is a questionnaire consisting of 10 questions. The total score ranges from 10 to 50 (higher score indicate worst quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: KPEK FKUI-RSCM, Principal Investigator — The Health Research Ethics Commitee - Faculty of Medicine Universitas Indonesia and Dr. Cipto Mangunkusumo National Hospital
Locations (1):
- Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No